CLINICAL TRIAL: NCT03595176
Title: Prospective, Multicenter, Single-Arm, Global IDE Study of the Shockwave Coronary Intravascular Lithotripsy (IVL) System With the Shockwave C2 Coronary IVL Catheter in Calcified Coronary Arteries
Brief Title: Disrupt CAD III With the Shockwave Coronary IVL System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 61982
Record Dates: First submitted 2018-06-22; First posted 2018-07-23 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Intravascular Lithotripsy; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Lithotripsy

STUDY DESIGN:
Intervention Model Description: The Coronary IVL System is a proprietary balloon catheter system designed to enhance stent outcomes by enabling delivery of the calcium disrupting capability of lithotripsy prior to balloon dilatation at low pressures. The Coronary IVL System consists of an IVL Balloon Catheter with two integrated pairs of lithotripsy emitters, a Lithotripsy Generator, and Connector Cable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Coronary Lithotripsy System (Experimental): All subjects will receive lithotripsy treatment from the Shockwave Medical Coronary IVL System
  Interventions: Device: Lithotripsy

INTERVENTIONS:
Device: Lithotripsy — Deliver Lithotripsy to the target vessel prior to placing a coronary stent.

SUMMARY:
The study design is a prospective, multicenter, single-arm, global IDE study to evaluate the safety and effectiveness of the Shockwave Medical Coronary Intravascular Lithotripsy (IVL) System in de novo, calcified, stenotic coronary arteries prior to stenting. Disrupt CAD III is being conducted as a staged pivotal study.

DETAILED DESCRIPTION:
Subject Population: Subjects ≥ 18 years of age with de novo, calcified coronary artery lesions presenting with stable, unstable or silent ischemia that are suitable for percutaneous coronary intervention (PCI). Approximately 392 subjects at 50 sites will be enrolled. A minimum of 50% of the total enrollment will come from the United States.Subjects will be followed through discharge, 30 days, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI
3. For patients with unstable ischemic heart disease, biomarkers (troponin or CK-MB) must be less than or equal to the upper limit of lab normal within 12 hours prior to the procedure (note: if both labs are drawn, both must be normal).
4. For patients with stable ischemic heart disease, biomarkers may be drawn prior to the procedure or at the time of the procedure from the side port of the sheath.

   1. If drawn prior to the procedure, biomarkers (troponin or CK-MB) must be less than or equal to the upper limit of lab normal within 12 hours of the procedure (note: if both labs are drawn, both must be normal).
   2. If biomarkers are drawn at the time of the procedure from the side port of the sheath prior to any intervention, biomarker results do not need to be analyzed prior to enrollment (note: CK-MB is required if drawn from the sheath).
5. Left ventricular ejection fraction >25% within 6 months (note: in the case of multiple assessments of LVEF, the measurement closest to enrollment will be used for this criteria; may be assessed at time of index procedure)
6. Subject or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures
7. Lesions in non-target vessels requiring PCI may be treated either:

   1. >30 days prior to the study procedure if the procedure was unsuccessful or complicated; or
   2. >24 hours prior to the study procedure if the procedure was successful and uncomplicated (defined as a final lesion angiographic diameter stenosis <30% and TIMI 3 flow (visually assessed) for all non-target lesions and vessels without perforation, cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation, and with no post-procedure biomarker elevation >normal; or
   3. >30 days after the study procedure

   Angiographic Inclusion Criteria
8. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
9. Single de novo target lesion stenosis of protected LMCA, or LAD, RCA or LCX (or of their branches) with:

   1. Stenosis of ≥70% and <100% or
   2. Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80, or iFR <0.90 or IVUS or OCT minimum lumen area ≤4.0 mm²
10. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm
11. The lesion length must not exceed 40 mm
12. The target vessel must have TIMI flow 3 at baseline (visually assessed; may be assessed after pre- dilatation)
13. Evidence of calcification at the lesion site by, a) angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, OR by b) IVUS or OCT, with presence of ≥270 degrees of calcium on at least 1 cross section
14. Ability to pass a 0.014" guide wire across the lesion

Exclusion Criteria:

1. Any comorbidity or condition which may reduce compliance with this protocol, including follow-up visits
2. Subject is a member of a vulnerable population as defined in 21 CFR 56.111, including individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention
3. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint
4. Subject is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment)
5. Unable to tolerate dual antiplatelet therapy (i.e., aspirin, and either clopidogrel, prasugrel, or ticagrelor) for at least 6 months (for patients not on oral anticoagulation)
6. Subject has an allergy to imaging contrast media which cannot be adequately pre-medicated
7. Subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure, defined as a clinical syndrome consistent with an acute coronary syndrome with troponin or CK-MB greater than 1 times the local laboratory's upper limit of normal
8. New York Heart Association (NYHA) class III or IV heart failure
9. Renal failure with serum creatinine >2.5 mg/dL or chronic dialysis
10. History of a stroke or transient ischemic attack (TIA) within 6 months, or any prior intracranial hemorrhage or permanent neurologic deficit
11. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months
12. Untreated pre-procedural hemoglobin <10 g/dL or intention to refuse blood transfusions if one should become necessary
13. Coagulopathy, including but not limited to platelet count <100,000 or International Normalized ratio (INR) > 1.7 (INR is only required in subjects who have taken warfarin within 2 weeks of enrollment)
14. Subject has a hypercoagulable disorder such as polycythemia vera, platelet count >750,000 or other disorders
15. Uncontrolled diabetes defined as a HbA1c greater than or equal to 10%
16. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics
17. Subjects in cardiogenic shock or with clinical evidence of left-sided heart failure (S3 gallop, pulmonary rales, oliguria, or hypoxemia)
18. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
19. Subjects with a life expectancy of less than 1 year
20. Non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days prior to the index procedure
21. Planned non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days after the index procedure
22. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
23. Planned use of atherectomy, scoring or cutting balloon, or any investigational device other than lithotripsy
24. High SYNTAX Score (≥33) if assessed as standard of care, unless the local heart team has met and recommends PCI is the most appropriate treatment for the patient
25. Unprotected left main diameter stenosis >30%
26. Target vessel is excessively tortuous defined as the presence of two or more bends >90º or three or more bends >75º
27. Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel
28. Evidence of aneurysm in target vessel within 10 mm of the target lesion
29. Target lesion is an ostial location (LAD, LCX, or RCA, within 5 mm of ostium) or an unprotected left main lesion
30. Target lesion is a bifurcation with ostial diameter stenosis ≥30%
31. Second lesion with >50% stenosis in the same target vessel as the target lesion including its side branches
32. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
33. Previous stent within the target vessel implanted within the last year
34. Previous stent within 10 mm of the target lesion regardless of the timing of its implantation
35. Angiographic evidence of a dissection in the target vessel at baseline or after guidewire passage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2022-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD,FACC,FSCAI, Study Chair — The Christ Hospital Heart and Vascular Center and The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital; Gregg W Stone, MD,FACC,FSCAI, Study Chair — Columbia University; Jonathan Hill, MD, Study Chair — Royal Brompton and Harefield NHS Foundation Trust
Locations (48):
- United States (39):
  - Honor Health, Scottsdale, Arizona
  - Scripps Clinic, La Jolla, California
  - University of California, San Diego (UCSD) - Medical Center, La Jolla, California
  - St. Joseph Hospital, Orange, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Advocate Health and Hospitals Corporation - Edward Hospital, Oakbrook Terrace, Illinois
  - St. Vincent Heart Center of Indiana, LLC, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - New York University (NYU) Langone Medical Center, New York, New York
  - Columbia University Medical Center/ New York Presbyterian, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Durham VA Health Care System, Durham, North Carolina
  - NC Heart and Vascular, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute Inc., Wormleysburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
  - Charleston Area Medical Center (CAMC) - Health Education & Research Institute, Charleston, West Virginia
- France (3):
  - Clinique Pasteur, Toulouse, Cedex 3
  - Clinique des Domes - Pole Sante Republique, Clermont-Ferrand
  - Institute Cardiovasculaire Paris Sud, Massy
- Germany (3):
  - Universitaetsklinikum Giessen and Marburg GmbH, Marburg, CET
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Rheinland Klinikum Neuss GmbH - Lukaskrankenhaus Neuss, Neuss
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank
  - St. Bartholomew's Hospital, London
  - King's College Hospital, London

REFERENCES:
- [Result] Hill JM, Kereiakes DJ, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease. J Am Coll Cardiol. 2020 Dec 1;76(22):2635-2646. doi: 10.1016/j.jacc.2020.09.603. Epub 2020 Oct 15. PMID 33069849
- [Result] Kereiakes DJ, Hill JM, Ben-Yehuda O, Maehara A, Alexander B, Stone GW. Evaluation of safety and efficacy of coronary intravascular lithotripsy for treatment of severely calcified coronary stenoses: Design and rationale for the Disrupt CAD III trial. Am Heart J. 2020 Jul;225:10-18. doi: 10.1016/j.ahj.2020.04.005. Epub 2020 Apr 18. PMID 32470635
- [Derived] Kereiakes DJ, Di Mario C, Riley RF, Fajadet J, Shlofmitz RA, Saito S, Ali ZA, Klein AJ, Price MJ, Hill JM, Stone GW. Intravascular Lithotripsy for Treatment of Calcified Coronary Lesions: Patient-Level Pooled Analysis of the Disrupt CAD Studies. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1337-1348. doi: 10.1016/j.jcin.2021.04.015. Epub 2021 May 3. PMID 33939604
- See also: Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Lesions: 1-Year Results From the Disrupt CAD III Study — https://doi.org/10.1016/j.jscai.2021.100001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment and enrollment took place at 47 global centers including 38 in the United States and 9 in Europe between January 9, 2019 and March 27, 2020. A total of 431 subjects with de novo, calcified, stenotic, coronary arteries were enrolled and treated with the Coronary Intravascular Lithotripsy (IVL) System.
Pre-assignment Details: 431 subjects were enrolled into the study. The definition of enrollment is when the subject signs informed consent, meets all inclusion criteria, none of the exclusion criteria, and the IVL catheter has been inserted over a 0.014 guidewire which had been previously passed across the study lesion.
Groups:
- Coronary IVL System (Roll-In): The first subject enrolled at each site is considered a roll-in. Per protocol, data on roll-in subjects were collected through 30 days, at which time subject participation was complete.
- Coronary IVL System (Pivotal): The pivotal analysis set was the primary analysis cohort used to assess the primary safety and effectiveness endpoints. Data on pivotal subjects was collected through 30 days for primary endpoints. Long-term follow-up for pivotal subjects to 24 months is complete.
Period: Overall Study
Arm/Group | Coronary IVL System (Roll-In) | Coronary IVL System (Pivotal)
Started | 47 | 384
Completed | 47 | 381
Not Completed | 0 | 3
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coronary IVL System (Roll-In) | Coronary IVL System (Pivotal) | Total
Number analyzed (Participants) | 47 | 384 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (7.6) | 71.2 (8.6) | 71.1 (8.5)
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Median (Q1, Q3) | 72.0 [64.0 to 76.0] | 71.0 [66.0 to 77.0] | 71.0 [66.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 90 | 102
  Male | 35 | 294 | 329
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 16 | 17
  Not Hispanic or Latino | 41 | 330 | 371
  Unknown or Not Reported | 5 | 38 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 13 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 12 | 15
  White | 35 | 318 | 353
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 38 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 335 | 373
  Europe | 9 | 49 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Freedom From Major Adverse Cardiac Events (MACE) Within 30 Days Post-procedure
Description: The primary safety endpoint was freedom from MACE at 30 days - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR). The primary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: Data collected from the roll-in subjects were not pre-specified to be reported as a Primary Outcome Measure; therefore, only pivotal group is reported. Additionally, one subject was excluded from the primary safety endpoint analysis due to insufficient follow-up (<23 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 383
percentage of participants | 92.2 [89.9 to NA] — The hypothesis test was a one-sided asymptotic Wald (normal approximation-based) confidence interval for a binomial proportion against a performance goal.

2. Primary Outcome: Number of Participants With Procedural Success (Residual Stenosis <50%)
Description: The primary effectiveness endpoint was Procedural Success defined as stent delivery with a residual in-stent stenosis <50% (core laboratory assessed) and without in-hospital MACE. The primary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 6 hours post procedure
Population: Data collected from the roll-in subjects were not pre-specified to be reported as a Primary Outcome Measure; therefore, only pivotal group is reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 92.4 [90.2 to NA] — The hypothesis test was a one-sided asymptotic Wald (normal approximation-based) confidence interval for a binomial proportion against a performance goal.

3. Secondary Outcome: Number of Participants With Device Crossing Success
Description: Device Crossing Success defined as the ability to deliver the IVL catheter across the target lesion, and delivery of lithotripsy without serious angiographic complications immediately after IVL. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: at end of procedure
Population: Data collected from the roll-in subjects were not pre-specified to be reported as a Secondary Outcome Measure; therefore, only pivotal group is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
Participants | 368

4. Secondary Outcome: Number of Participants With Angiographic Success (Residual Stenosis <50%)
Description: Angiographic Success defined as stent delivery with <50% residual stenosis and without serious angiographic complications. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: at end of procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
Participants | 370

5. Secondary Outcome: Number of Participants With Procedural Success (Residual Stenosis <=30%)
Description: Procedural Success defined as stent delivery with a residual stenosis <=30% (core laboratory assessed) and without in-hospital MACE. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 6 hours post procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
Participants | 354

6. Secondary Outcome: Number of Participants With Angiographic Success (Residual Stenosis <=30%)
Description: Angiographic Success defined as stent delivery with <=30% residual stenosis and without serious angiographic complications. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: at end of procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
Participants | 369

7. Secondary Outcome: Number of Participants With Serious Angiographic Complications
Description: Serious Angiographic Complications defined as severe dissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: at end of procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
Participants | 12

8. Secondary Outcome: MACE Rate at 6 Months
Description: MACE at 6 months - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR) - is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 10.2

9. Secondary Outcome: MACE Rate at 12 Months
Description: MACE at 12 months - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR) - is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 13.6

10. Secondary Outcome: MACE Rate at 24 Months
Description: MACE at 24 months - a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR) - is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 18.9

11. Secondary Outcome: Target Lesion Failure (TLF) Rate at 30 Days
Description: Target lesion failure (TLF) is defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods. 30 day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.6

12. Secondary Outcome: Target Lesion Failure (TLF) Rate at 6 Months
Description: TLF is defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods. For 6 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 9.1

13. Secondary Outcome: Target Lesion Failure (TLF) Rate at 12 Months
Description: TLF is defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods. For 12 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 11.9

14. Secondary Outcome: Target Lesion Failure (TLF) Rate at 24 Months
Description: TLF is defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods. For 24 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 16.1

15. Secondary Outcome: All-Cause Death Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0.5

16. Secondary Outcome: All-Cause Death Rate at 6 Months
Description: All-cause death at 6 months is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.3

17. Secondary Outcome: All-Cause Death Rate at 12 Months
Description: All-cause death at 12 months is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.8

18. Secondary Outcome: All-Cause Death Rate at 24 Months
Description: All-cause death at 24 months is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 5.9

19. Secondary Outcome: Cardiac Death Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0.5

20. Secondary Outcome: Cardiac Death Rate at 6 Months
Description: Cardiac death at 6 months is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0.8

21. Secondary Outcome: Cardiac Death Rate at 12 Months
Description: Cardiac death at 12 months is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.1

22. Secondary Outcome: Cardiac Death Rate at 24 Months
Description: Cardiac death at 24 months is presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.7

23. Secondary Outcome: MI Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.3

24. Secondary Outcome: MI Rate at 6 Months
Description: MI is presented as a Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 9.1

25. Secondary Outcome: MI Rate at 12 Months
Description: MI is presented as a Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 10.5

26. Secondary Outcome: MI Rate at 24 Months
Description: MI is presented as a Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 12.6

27. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.3

28. Secondary Outcome: TV-MI Rate at 6 Months
Description: TV-MI is presented as a Kaplan-Meier estimated event rate at 6 months. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.6

29. Secondary Outcome: TV-MI Rate at 12 Months
Description: TV-MI is presented as a Kaplan-Meier estimated event rate at 12 months. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.8

30. Secondary Outcome: TV-MI Rate at 24 Months
Description: TV-MI is presented as a Kaplan-Meier estimated event rate at 24 months. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 8.1

31. Secondary Outcome: Procedural MI Rate at 30 Days
Description: Periprocedural MI defined as CK-MB > 3x upper limit of lab normal (ULN). 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 6.8

32. Secondary Outcome: Procedural MI Rate at 6 Months
Description: Periprocedural MI defined as CK-MB > 3x upper limit of lab normal (ULN). For 6 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 6.8

33. Secondary Outcome: Procedural MI Rate at 12 Months
Description: Periprocedural MI defined as CK-MB > 3x upper limit of lab normal (ULN). For 12 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 6.8

34. Secondary Outcome: Procedural MI Rate at 24 Months
Description: Periprocedural MI defined as CK-MB > 3x upper limit of lab normal (ULN). For 24 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 6.8

35. Secondary Outcome: Non-Procedural MI Rate at 30 Days
Description: Non-Procedural MI defined as spontaneous MI beyond discharge (4th Universal Definition). 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.0

36. Secondary Outcome: Non-Procedural MI Rate at 6 Months
Description: Non-Procedural MI defined as spontaneous MI beyond discharge (4th Universal Definition). For 6 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 3.2

37. Secondary Outcome: Non-Procedural MI Rate at 12 Months
Description: Non-Procedural MI defined as spontaneous MI beyond discharge (4th Universal Definition). For 12 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 4.8

38. Secondary Outcome: Non-Procedural MI Rate at 24 Months
Description: Non-Procedural MI defined as spontaneous MI beyond discharge (4th Universal Definition). For 24 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.2

39. Secondary Outcome: Ischemia-Driven Target Vessel Revascularization (ID-TVR) Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.6

40. Secondary Outcome: ID-TVR Rate at 6 Months
Description: For 6 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.9

41. Secondary Outcome: ID-TVR Rate at 12 Months
Description: For 12 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 6.0

42. Secondary Outcome: ID-TVR Rate at 24 Months
Description: For 24 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 8.5

43. Secondary Outcome: Ischemia-Driven Target Lesion Revascularization (ID-TLR) Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.3

44. Secondary Outcome: ID-TLR Rate at 6 Months
Description: as for outcome 40
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.4

45. Secondary Outcome: ID-TLR Rate at 12 Months
Description: as for outcome 41
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 4.3

46. Secondary Outcome: ID-TLR Rate at 24 Months
Description: as for outcome 42
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 6.4

47. Secondary Outcome: Non-ID-TVR Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

48. Secondary Outcome: Non-ID-TVR Rate at 6 Months
Description: as for outcome 40
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

49. Secondary Outcome: Non-ID-TVR Rate at 12 Months
Description: as for outcome 41
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

50. Secondary Outcome: Non-ID-TVR Rate at 24 Months
Description: as for outcome 42
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

51. Secondary Outcome: Non-ID-TLR Rate at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

52. Secondary Outcome: Non-ID-TLR Rate at 6 Months
Description: as for outcome 40
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

53. Secondary Outcome: Non-ID-TLR Rate at 12 Months
Description: as for outcome 41
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

54. Secondary Outcome: Non-ID-TLR Rate at 24 Months
Description: as for outcome 42
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0

55. Secondary Outcome: Any Revascularizations Rate at 30 Days
Description: Any revascularizations (ID and non-ID) at 30 days. 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.6

56. Secondary Outcome: Any Revascularizations Rate at 6 Months
Description: Any revascularizations (ID and non-ID) at 6 months, presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.9

57. Secondary Outcome: Any Revascularizations Rate at 12 Months
Description: Any revascularizations (ID and non-ID) at 12 months, presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 12.3

58. Secondary Outcome: Any Revascularizations Rate at 24 Months
Description: Any revascularizations (ID and non-ID) at 24 months, presented as a Kaplan-Meier estimated event rate. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 15.4

59. Secondary Outcome: Stent Thrombosis Rate at 30 Days
Description: Any stent thrombosis (definite, probable, definite or probable) according to Academic Research Consortium (ARC) criteria, as referenced from Cutlip, D.E. et al. Clinical End Points in Coronary Stent Trials. Circ. 2007.115.2344-51. 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 0.8

60. Secondary Outcome: Stent Thrombosis Rate at 6 Months
Description: Any stent thrombosis (definite, probable, definite or probable) according to Academic Research Consortium (ARC) criteria, as referenced from Cutlip, D.E. et al. Clinical End Points in Coronary Stent Trials. Circ. 2007.115.2344-51. For 6 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.3

61. Secondary Outcome: Stent Thrombosis Rate at 12 Months
Description: Any stent thrombosis (definite, probable, definite or probable) according to Academic Research Consortium (ARC) criteria, as referenced from Cutlip, D.E. et al. Clinical End Points in Coronary Stent Trials. Circ. 2007.115.2344-51. For 12 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 1.6

62. Secondary Outcome: Stent Thrombosis Rate at 24 Months
Description: Any stent thrombosis (definite, probable, definite or probable) according to Academic Research Consortium (ARC) criteria, as referenced from Cutlip, D.E. et al. Clinical End Points in Coronary Stent Trials. Circ. 2007.115.2344-51. For 24 months, rates are presented as Kaplan-Meier estimated event rates. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.7

63. Secondary Outcome: Rate of MI Using the 4th Universal Definition at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.3

64. Secondary Outcome: Rate of MI Using the 4th Universal Definition at 6 Months
Description: as for outcome 40
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.3

65. Secondary Outcome: Rate of MI Using the 4th Universal Definition at 12 Months
Description: as for outcome 41
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.3

66. Secondary Outcome: Rate of MI Using the 4th Universal Definition at 24 Months
Description: as for outcome 42
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 7.3

67. Secondary Outcome: Rate of MI Using the Society for Cardiovascular Angiography and Interventions (SCAI) Definition at 30 Days
Description: 30-day rates are presented as proportions. The secondary endpoints were analyzed using the Pivotal Analysis Set.
Time Frame: within 30 days of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.6

68. Secondary Outcome: Rate of MI Using the SCAI Definition at 6 Months
Description: as for outcome 40
Time Frame: within 6 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.6

69. Secondary Outcome: Rate of MI Using the SCAI Definition at 12 Months
Description: as for outcome 41
Time Frame: within 12 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.6

70. Secondary Outcome: Rate of MI Using the SCAI Definition at 24 Months
Description: as for outcome 42
Time Frame: within 24 months of index procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Coronary IVL System (Pivotal)
Number analyzed (Participants) | 384
percentage of participants | 2.6

ADVERSE EVENTS:
Time Frame: within 30 days of index procedure for both Roll-In and Pivotal arms, and through 24 months for Pivotal arm only
Description: Long-term follow-up for pivotal subjects to 24 months is complete.
Groups:
- Coronary IVL System (Roll-In) Through 30 Days: Adverse events reported through 30 days post-procedure for Roll-In subjects. The first subject enrolled at each site is considered a roll-in. Per protocol, data on roll-in subjects were collected through 30 days, at which time subject participation was complete.
- Coronary IVL System (Pivotal) Through 30 Days: Adverse events reported through 30 days post-procedure for Pivotal subjects. The pivotal analysis set was the primary analysis cohort used to assess the primary safety and effectiveness endpoints.
- Coronary IVL System (Pivotal) Through 12 Months: Adverse events reported through 12 months post-procedure for Pivotal subjects. Adverse event data on pivotal subjects was collected through 12 months for long-term follow-up.
- Coronary IVL System (Pivotal) Through 24 Months: Adverse events reported through 24 months post-procedure for Pivotal subjects. Adverse event data on pivotal subjects was collected through 24 months for long-term follow-up.
Arm/Group | Coronary IVL System (Roll-In) Through 30 Days | Coronary IVL System (Pivotal) Through 30 Days | Coronary IVL System (Pivotal) Through 12 Months | Coronary IVL System (Pivotal) Through 24 Months
All-Cause Mortality (participants affected / at risk) | 0/47 | 2/384 | 7/384 | 22/384
Serious Adverse Events (participants affected / at risk) | 4/47 | 54/384 | 136/384 | 173/384
Other Adverse Events (participants affected / at risk) | 15/47 | 54/384 | 140/384 | 162/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary IVL System (Roll-In) Through 30 Days (N=47) | Coronary IVL System (Pivotal) Through 30 Days (N=384) | Coronary IVL System (Pivotal) Through 12 Months (N=384) | Coronary IVL System (Pivotal) Through 24 Months (N=384)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5) | 5 (5)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 11 (11) | 11 (11) | 11 (11)
Myocardial infarction (Cardiac disorders) | 0 (0) | 8 (10) | 16 (18) | 24 (27)
Arrhythmia (Cardiac disorders) | 0 (0) | 6 (10) | 15 (20) | 19 (26)
Angina pectoris (Cardiac disorders) | 0 (0) | 5 (5) | 15 (21) | 17 (23)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (8)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 4 (5) | 4 (5)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 5 (5) | 8 (9) | 9 (10)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 6 (6) | 11 (11)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myocardial necrosis marker increased (elevated cardiac biomarker) (Investigations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) — Cardiac biomarker includes troponin or CK-MB
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (6)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (3) | 3 (6)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 4 (4) | 8 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 10 (11) | 15 (17)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (5)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Shock (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 4 (4) | 6 (6)
Plaque shift (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 5 (7)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 14 (15) | 24 (26)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Vascular access site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (7)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug withdrawal convulsions (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (6) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nomocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eccrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary IVL System (Roll-In) Through 30 Days (N=47) | Coronary IVL System (Pivotal) Through 30 Days (N=384) | Coronary IVL System (Pivotal) Through 12 Months (N=384) | Coronary IVL System (Pivotal) Through 24 Months (N=384)
Myocardial necrosis marker increased (elevated cardiac biomarker) (Investigations) | 10 (12) | 54 (60) | 57 (64) | 58 (66) — Cardiac biomarker includes troponin or CK-MB
Angina pectoris (Cardiac disorders) | 3 (3) | 17 (18) | 37 (40) | 43 (52) — Pivotal group through 30 days does not meet 5% frequency threshold for reporting
Coronary artery dissection (Cardiac disorders) | 3 (3) | 18 (18) | 18 (18) | 18 (18) — Pivotal group does not meet 5% frequency threshold for reporting
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 16 (18) | 32 (38) | 34 (42) — Roll-in and pivotal groups through 30 days do not meet 5% frequency threshold for reporting
Arrhythmia (Cardiac disorders) | 0 (0) | 7 (8) | 25 (26) | 29 (34) — Roll-in and pivotal groups through 30 days do not meet 5% frequency threshold for reporting
Infection (Infections and infestations) | 1 (1) | 1 (1) | 25 (27) | 30 (34) — Roll-in and pivotal groups through 30 days do not meet 5% frequency threshold for reporting
Non-cardiac chest pain (General disorders) | 0 (0) | 10 (11) | 19 (21) | 23 (27) — Roll-in and pivotal groups through 30 days and 12 months do not meet 5% frequency threshold for reporting
Fatigue (General disorders) | 2 (2) | 4 (4) | 14 (14) | 21 (22) — Roll-in and pivotal groups through 30 days and 12 months do not meet 5% frequency threshold for reporting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03595176/Prot_SAP_001.pdf